CLINICAL TRIAL: NCT03980470
Title: Usefulness of Deep-Learning Image Reconstruction for Cardiac Computed Tomography Angiography - a Prospective, Non-randomized Observational Trial
Brief Title: Deep-Learning Image Reconstruction in CCTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Ronny R Buechel, MD, PD Dr. med. Ronny R. Buechel, University of Zurich
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: USZ-2019-00533
Record Dates: First submitted 2019-05-24; First posted 2019-06-10 (Actual); Results first posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-10

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Normal-dose versus Low-dose (Other): The standard intervention consists of the routinely performed cardiac CT datasets reconstructed with a standard iterative reconstruction algorithm (ASIR-V). Median radiation dose is about 0.5 mSv, range between about 0.2 and 1.2 mSv; median contrast agent administration about 45 mL, range between 35 and 55 mL.
  The experimental intervention is an additional CT scan with a lower dose (about 20 to 50% decrease) and a similar contrast agent administration that is reconstructed with a deep-learning image reconstruction immediately after the clinical CT scan. The additional time required is about 5 minutes.
  Interventions: Device: TrueFidelity

INTERVENTIONS:
Device: TrueFidelity — TrueFidelity (Deep Learning Image Reconstruction, DLIR) software by GE Healthcare.
  The medical device in question is a novel reconstruction algorithm for raw CT data which is based on artificial intelligence approaches, namely deep-learning iterative reconstruction (DLIR). This DLIR algorithm will be installed on the console of the CT Revolution scanning device, which is in routine clinical use for cardiac CT scans at the Department of Nuclear Medicine at the University Hospital Zurich. Purpose of this installation is the assessment of the performance of the DLIR algorithm during a limited time span of six weeks.
  The algorithm will be CE-marked at the time of installation and use (statement by GE Healthcare provided separately). Its intended use is the reconstruction of CT datasets.
  Of note, the novel DLIR algorithm will not substitute any clinical routine procedures currently in use. That is, diagnosis will still be made using the standard reconstruction algorithms.

SUMMARY:
Cardiac CT allows the assessment of the heart and of the coronary arteries by use of ionising radiation. Although radiation exposure was significantly reduced in recent years, further decrease in radiation exposure is limited by increased image noise and deterioration in image quality. Recent evidence suggests that further technological refinements with artificial intelligence allows improved post-processing of images with reduction of image noise.

The present study aims at assessing the potential of a deep-learning image reconstruction algorithm in a clinical setting. Specifically, after a standard clinical scan, patients are scanned with lower radiation exposure and reconstructed with the DLIR algorithm. This interventional scan is then compared to the standard clinical scan.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for cardiac CT angiography
* Age ≥ 18 years
* Written informed consent

Exclusion Criteria:

* Pregnancy or breast-feeding
* Enrollment of the investigator, his/her family members, employees and other dependent persons
* Renal insufficiency (GFR below 35 mL/min/1.73 m²)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-05-08 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronny R Buechel, MD, Principal Investigator — Director of Cardiac Imaging
Locations (1):
- University Hospital, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benz DC, Grani C, Hirt Moch B, Mikulicic F, Vontobel J, Fuchs TA, Stehli J, Clerc OF, Possner M, Pazhenkottil AP, Gaemperli O, Buechel RR, Kaufmann PA. Minimized Radiation and Contrast Agent Exposure for Coronary Computed Tomography Angiography: First Clinical Experience on a Latest Generation 256-slice Scanner. Acad Radiol. 2016 Aug;23(8):1008-14. doi: 10.1016/j.acra.2016.03.015. Epub 2016 May 9. PMID 27174030
- [Background] Benz DC, Fuchs TA, Grani C, Studer Bruengger AA, Clerc OF, Mikulicic F, Messerli M, Stehli J, Possner M, Pazhenkottil AP, Gaemperli O, Kaufmann PA, Buechel RR. Head-to-head comparison of adaptive statistical and model-based iterative reconstruction algorithms for submillisievert coronary CT angiography. Eur Heart J Cardiovasc Imaging. 2018 Feb 1;19(2):193-198. doi: 10.1093/ehjci/jex008. PMID 28200212
- [Background] Sahiner B, Pezeshk A, Hadjiiski LM, Wang X, Drukker K, Cha KH, Summers RM, Giger ML. Deep learning in medical imaging and radiation therapy. Med Phys. 2019 Jan;46(1):e1-e36. doi: 10.1002/mp.13264. Epub 2018 Nov 20. PMID 30367497
- [Background] Toprak O. Conflicting and new risk factors for contrast induced nephropathy. J Urol. 2007 Dec;178(6):2277-83. doi: 10.1016/j.juro.2007.08.054. Epub 2007 Oct 22. PMID 17936812
- [Background] Benz DC, Grani C, Hirt Moch B, Mikulicic F, Vontobel J, Fuchs TA, Stehli J, Clerc OF, Possner M, Pazhenkottil AP, Gaemperli O, Buechel RR, Kaufmann PA. A low-dose and an ultra-low-dose contrast agent protocol for coronary CT angiography in a clinical setting: quantitative and qualitative comparison to a standard dose protocol. Br J Radiol. 2017 Jun;90(1074):20160933. doi: 10.1259/bjr.20160933. Epub 2017 May 25. PMID 28406318

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: 08/May/2019 until 20/June/2019 Location: University Hospital Zurich, Department of Nuclear Medicine, Switzerland
Period: Overall Study
Arm/Group | Normal-dose Versus Low-dose
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Normal-dose Versus Low-dose
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 43
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 50
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Switzerland | 50

OUTCOME MEASURES:

1. Primary Outcome: Subjective Image Quality
Description: Subjective image quality as measured by Likert scale from 1 (non-evaluable) to 5 (excellent)
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: Score on a Likert scale (0-5) 5=best
Arm/Group | Normal-dose Versus Low-dose
Number analyzed (Participants) | 50
Score on a Likert scale (0-5) 5=best
  Low-Dose | 5 (0)
  Normal-Dose | 5 (0)

2. Secondary Outcome: Signal Intensity
Description: Signal intensity as average hounsfield units within a region of interest in the aortic root, change from experimental interventional to the control intervention
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: Hounsfield units
Arm/Group | Normal-dose Versus Low-dose
Number analyzed (Participants) | 50
Hounsfield units
  Low-Dose | 462 (76)
  Normal Dose | 443 (85)
Statistical Analysis 1: Comparison: Normal-dose Versus Low-dose; Test type: Superiority; p = 0.198, ANOVA

3. Secondary Outcome: Image Noise
Description: Image noise as standard deviation of hounsfield units within a region of interest in the aortic root, change from experimental interventional to the control intervention
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: Hounsfield units
Groups:
- Low-dose: The standard intervention consists of the routinely performed cardiac CT datasets reconstructed with a standard iterative reconstruction algorithm (ASIR-V). Median radiation dose is about 0.5 mSv, range between about 0.2 and 1.2 mSv; median contrast agent administration about 45 mL, range between 35 and 55 mL.
  The experimental intervention is an additional CT scan with a lower dose (about 20 to 50% decrease) and a similar contrast agent administration that is reconstructed with a deep-learning image reconstruction immediately after the clinical CT scan. The additional time required is about 5 minutes.
Arm/Group | Low-dose
Number analyzed (Participants) | 50
Hounsfield units
  Low-Dose | 27 (4)
  Normal-Dose | 28 (6)
Statistical Analysis 1: Comparison: Low-dose; Test type: Superiority; p = 0.9, ANOVA

4. Secondary Outcome: Signal-to-noise Ratio
Description: Signal-to-noise ratio
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Low-dose
Number analyzed (Participants) | 50
Ratio
  Low-Dose | 17 (3)
  Normal-Dose | 16 (2)
Statistical Analysis 1: Comparison: Low-dose; Test type: Superiority; p = 0.8, ANOVA

5. Secondary Outcome: Dose-length Products
Description: Comparison of dose-length products
Time Frame: Day 1
Measure: Median (Inter-Quartile Range); unit: mGy*cm
Arm/Group | Normal-Dose Versus Low-dose
Number analyzed (Participants) | 50
mGy*cm
  Low-Dose | 31 [25 to 34]
  Normal-Dose | 52 [42 to 58]
Statistical Analysis 1: Comparison: Normal-Dose Versus Low-dose; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Plaque Volumes
Description: Quantitative analysis of coronary artery plaque volumes
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Normal-Dose Versus Low-dose
Number analyzed (Participants) | 50
mm^3
  Low-Dose | 12.42 (13.14)
  Normal-Dose | 13.84 (14.41)
Statistical Analysis 1: Comparison: Normal-Dose Versus Low-dose; Test type: Other — Bland-Altmann analysis (bias); Mean Difference (Final Values) = -1.42

ADVERSE EVENTS:
Time Frame: 1 day
Groups:
- Low-dose: The experimental intervention is an additional CT scan with a lower dose (about 20 to 50% decrease) and a similar contrast agent administration that is reconstructed with a deep-learning image reconstruction immediately after the clinical CT scan. The additional time required is about 5 minutes.
  TrueFidelity: TrueFidelity (Deep Learning Image Reconstruction, DLIR) software by GE Healthcare.
  The medical device in question is a novel reconstruction algorithm for raw CT data which is based on artificial intelligence approaches, namely deep-learning iterative reconstruction (DLIR). This DLIR algorithm will be installed on the console of the CT Revolution scanning device, which is in routine clinical use for cardiac CT scans at the Department of Nuclear Medicine at the University Hospital Zurich. Purpose of this installation is the assessment of the performance of the DLIR algorithm during a limited time span of six weeks.
  The algorithm will be CE-marked at the time of installation and use (statement by GE Healthcare provided separately). Its intended use is the reconstruction of CT datasets.
  Of note, the novel DLIR algorithm will not substitute any clinical routine procedures currently in use. That is, diagnosis will still be made using the standard reconstruction algorithms.
- Normal-dose: The control intervention consists of the routinely performed cardiac CT datasets reconstructed with a standard iterative reconstruction algorithm (ASIR-V). Median radiation dose is about 0.5 mSv, range between about 0.2 and 1.2 mSv; median contrast agent administration about 45 mL, range between 35 and 55 mL.
Arm/Group | Low-dose | Normal-dose
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-23): https://cdn.clinicaltrials.gov/large-docs/70/NCT03980470/Prot_SAP_000.pdf